CLINICAL TRIAL: NCT01704508
Title: Efficacy and Safety of Artemether + Lumefantrine and Dihydroartemisinin + Piperaquine for the Treatment of Uncomplicated Malaria in Guinea-Bissau.
Brief Title: Improving Anti-malarial Treatment Options in Guinea-Bissau - Part A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eurartesim-2012
Record Dates: First submitted 2012-10-09; First posted 2012-10-11 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2015-08

CONDITIONS: Malaria
Keywords: Falciparum malaria; children; treatment
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): 6-dose regime will be used:
  Interventions: Drug: Artemether-lumefantrine
- Dihydroartemisinin-piperaquine (Active Comparator): A 3 dose regime will be used
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine
  Other Names: Coartem (R)
  Arms: Artemether-lumefantrine
Drug: Dihydroartemisinin-piperaquine
  Other Names: Eurartesim
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Plasmodium falciparum causes malaria and approximately 665 000 deaths each year. chloroquine and sulphadoxine-pyrimethamine resistant P. falciparum are widespread. An artemisinin derivative combined with lumefantrine, amodiaquine or piperaquine is therefore recommended for the treatment of malaria in Africa. However, artemisinin resistance appears to be developing and resistance/tolerance to amodiaquine and lumefantrine exists. We are presently conducting a study in Guinea-Bissau. Preliminary data indicates that the effectiveness and availability of artemether-lumefantrine (AL), the 1st line drug, is poor. Consequently there is a need for another treatment option. Dihydroartemisinin-piperaquine (DP) has been shown to be efficacious and well tolerated in several African countries and is therefore such an option. A clinical trial comparing the safety and efficacy of artemether-lumefantrine and dihydroartemisinin-piperaquine is therefore needed.

Parents to children seeking Bandim Health Centre (CSB) with symptoms compatible with malaria will be informed of the study. If accepting and the child fulfil the inclusion criteria, the child will be randomised to treatment with either AL or DP. The treatment will be given supervised at the health centre in the morning and the evening on day 0, day 1, and day 2.

At each visit and in the morning on day 3, the child will be examined, the mother asked for any symptoms and signs of side-effects, the temperature measured. Furthermore, a blood sample will be taken for examination of malaria parasites. On day 0 samples for measurement of antimalarial drugs and for genotyping of the parasites will be taken on filterpaper. In a subgroup of 50 children a blood sample for in vitro culturing and for analysis of the number of leucocytes will also be taken.

After having finished the treatment the children will be followed on day 7 and then once a week until day 42. At each visit the condition of the child will be examined and a bloodsample taken for examination of parasites in the blood. Furthermore, a filterpaper bloodsample will be collected for measurement of the drug concentration of if the child has recrudescence for genotyping of the parasites. On day 0, 3 and 42 the haemoglobin level will be examined.

The result of the two treatments will be evaluated by comparing the number of children with recurrent parasitaemia, both corrected and uncorrected (recrudescence vs. reinfections). This will be presented as adequate clinical and parasitological response rates PCR-corrected and PCR-uncorrected. Furthermore, the chance in haemoglobin level from day 0 till day 3 and till day 42 will be compared. The concentration of the antimalarial drug in the blood samples taken at the visit before the re-parasitaemia will be capered to the concentrations in children without re-parasitaemia.

Assuming a 20% loss to follow up a total of 346 children should be included. For the children included, health care and medications at Bandim Health Centre will be free during the study period but no other gifts or payments will be made.

Results will be presented to the staff at the Bandim health centre and the ministry of Health and will be published in an international peer reviewed journal.

DETAILED DESCRIPTION:
Background Plasmodium falciparum causes malaria and approximately 665 000 deaths each year. Previously chloroquine (CQ) and sulphadoxine-pyrimethamine were the principle drugs for the treatment of malaria. Due to widespread resistance to these drugs1, the World Health Organization recommends that P. falciparum in Africa should be treated with artemisinin + amodiaquine, artemether + lumefantrine (AL) or dihydroartemisinin + piperaquine2 (DP). However, resistance to artemisinins appears to be developing3,4, resistance to amodiaquine exists2 and treatment with AL rapidly selects for parasites with increased tolerance (5 times higher inhibitory concentration) to lumefantrine5-7.

In Guinea-Bissau, CQ remained efficacious until replaced by AL. This is explained by the use of a unique well tolerated high dose treatment schedule 8-10. Since the introduction of AL in 2008, the number of children with malaria has increased manyfold in Bissau in contrast with other African countries. Our data suggests that this increase is due unavailability of AL, poorer than expected effectiveness of AL and to an increased use of the second-line drug quinine. Quinine is typically given for 3 instead of 7 days and has very poor efficacy when used thus11. To counter this Guinea-Bissau needs an alternative cheap and easily dosed 2nd line drug that can also be used when AL is not available or when funding for AL no longer exists.

Dihydroartemisinin+piperaquine is a safe and well tolerated artemisinin based combination12. DP is taken once daily and has been shown to be highly efficacious (>95%) in several African settings13,14. DP also protects from re-infection for longer than AL14. As such this is a drug that could become an attractive treatment option in Guinea-Bissau. It has however, never been used in the country.

Aim Conduct an efficacy study with artemether + lumefantrine and dihydroartemisinin + piperaquine

1. To measure the efficacy and safety of AL and DP in children aged 6 months to 12 years suffering from uncomplicated P. falciparum malaria.
2. To determine the capacity of each drug combination to protect against re-infection.
3. To differentiate recrudescence from re-infections using PCR based methods
4. To determine whole blood concentrations of lumefantrine and piperaquine the week before reparasitaemia
5. To determine haemoglobin values on days 0, 3 and 42
6. To determine differential white blood cell counts on days 0, 3, 7, 14 and 21
7. To determine genetic polymorphisms in P. falciparum causing reparasitaemia,
8. To culture parasites from 50 children for further characterisation of P. falciparum geno- and phenotypes.

   2. Methods Study design This will be an open label, randomized, non inferiority trial conducted at the Bandim health centre, Guinea-Bissau. Children with uncomplicated malaria who meet study inclusion criteria will be enrolled, randomised to treatment with either AL or DP, treated on site and monitored for 42 days. The follow up will consist of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. The proportion of children experiencing therapeutic failure during the follow-up period will be used to estimate the efficacy of the study drugs. PCR analysis will be used to distinguish between a true recrudescence due to treatment failure and episodes of re-infection.

   Study Site and population Children aged 6 months to 12 years with uncomplicated P. falciparum malaria that attend the Bandim health centre.

   Timing and duration of the study The study will start in November 2012 and continue until 350 children are included. If this is not achieved in one year the study will run for 2 years.

   Inclusion criteria A) Age ≥6 months, and <13 years. B) Mono-infection with P. falciparum detected by microscopy. C) Parasitemia of 1.000-200.000/µl asexual forms. D) Axillary temperature ≥37.5 ˚C or a history of fever within 24 hours. E) Ability to swallow oral medication.

   F) Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule. G) Informed consent from a parent or guardian

   Exclusion criteria A) Signs or symptoms of severe malaria including the following symptoms Prostration. Impaired consciousness. Respiratory distress. Repeated generalised convulsions (three or more per 24 hours or 2 witnessed seizures in 24 hours). Circulatory collapse. Abnormal bleeding. Jaundice. Haemoglobinuria (dark red/black urine). Severe anaemia (Haemoglobin <5g/dl). Hyperparasitaemia (>200.000/ µl asexual forms) B) Presence of general danger signs in children under 5 including the following Prostration. Respiratory distress. Haemoglobin <5g/dl. Two or more convulsions within 24 hours. Persistent vomiting C) Presence of severe malnutrition. D) Any evidence of chronic disease or acute infection other than malaria. E) Regular medication which may interfere with antimalarial pharmacokinetics. F) History of hypersensitivity reactions or contraindications to AL, DP or quinine.

   G) Domicile outside the study area.

   Loss to follow up If a child is not seen on the day of follow up the child will be sought at home on two consecutive days and if possible contacted by mobile phone. At each subsequent weekly follow up three new attempts to see the child will be made.

   3. Treatment Antimalarial treatment Treatment with AL will be given according to a 6-dose regime. Treatment with DP will be given according to a 3 dose regime. Tablets of AL (20 mg artemether and 120 mg lumefantrine) will be obtained from the manufacturer. Tablets of DP (Eurartesim®) with 160mg/20mg or 320mg/40mg obtained from Sigma-Tau.

   Block Randomization Identical slips of paper specifying treatment arm AL or DP will be put into an envelope. Each envelope will contain 20 slips from each group and children will randomly select one slip.

   Concomitant treatment and medication that should not be used Paracetamol will be used to treat fever. Iron and vitamin supplementation will be given if required. Prior treatment with an antimalarial drug will not be considered as exclusion criteria. Children taking any drug with antimalarial activity (including antibiotics such as tetracycline or azithromycin) during the study period will be withdrawn.

   Rescue treatment If children vomit twice, they will receive therapy with quinine intramuscularly and will be withdrawn from the study. Any child with signs of severe or complicated malaria will be treated according to recommendations of the attending nurse. If a child meets criteria for early treatment failure, he or she will receive parenteral quinine. If a child meets criteria for late treatment failure he or she will be re-treated with AL.

   4. Evaluation Criteria Efficacy and safety evaluation Treatment outcomes will be early treatment failure, late clinical failure, late parasitological failure or adequate clinical and parasitological response as defined by the WHO2.

   Safety end points The incidence of any adverse event including neutropenia will be documented. All children will be asked routinely about previous symptoms and about symptoms that have emerged since the previous follow up visit. When clinically indicated, children will be evaluated and treated appropriately. All adverse events will be recorded in the case record forms.

   Clinical evaluation All children will be evaluated by an attending study nurse and the examination will include a physical examination, body weight, body (axillary) temperature as shown in table 3

   Microscopic examination Two thick and thin blood films for parasite counts and species identification will be obtained as shown in table 3 and whenever a child returns to the Bandim health centre. Slides will be stained using freshly prepared Giemsa and examined with 1000 x magnification. The number of asexual parasites per 200 white blood cells will be counted or, if parasitaemia is high, the number of white blood cells per 500 parasites will be counted. Parasite density will be assessed independently by 2 qualified microscopists. Discordant results will be read a third time.

   Genotyping, antimalarial drug concentration, haemoglobin and white blood cell count 100µL of blood will be collected on Whatman 3MM filter-paper using a capillary tube on day 0, 7, 14, 21, 28, 35, 42 and whenever reparasitaemia is detected. Filter-papers will be dried and then placed inside separate sealed plastic bags. Filter-papers and bags will be labelled with study number date and follow up day. The samples will be stored at -20˚C. Blood samples will be obtained at the same time that blood is taken for microscopy.

   In order to differentiate recrudescence from a re-infection genotyping using sequential analysis of pfglurp, pfmsp1 and pfmsp2 will be done21.

   The proportion of resistance associated genotypes in resistance associated genes including pfcrt, pfmdr1, pfmrp1 and pfcmu will be determined. Genotyping will be done at Karolinska Institutet, Stockholm, Sweden and/or Universidade do Minho, Portugal.

   Drug concentrations will be assessed on the week prior to reparasitaemia at Mahidol University Bangkok using high performance liquid chromatography (HPLC).

   Haemoglobin concentration will be determined on day 0, 3 and 42 using a haemocueTM At the same time that blood sampling for microscopy is done on Day 0, exactly 200μL of blood will also be taken for in vitro culturing from 50 patients. The blood will be put into medium and grown in vitro in an incubator at 37 ˚C. When a culture is established it will be frozen in liquid nitrogen for transport to Sweden or Portugal where extensive drug assays will be carried out.

   5. Study Assessment Screening and enrolment As part of the routine medical services provided at the health centre, all children with symptoms suggestive of malaria will be screened for malaria using a rapid diagnostic test. Positive tests are confirmed by microscopy. Children fulfilling inclusion critera will be invited to participate in the study following informed consent.

   Follow up Children will be given a unique personal identification number and be given treatment after informed consent. The basic follow up schedule is shown below. Treatments, information to the children, clinical observations and adverse events will be recorded in the clinical record forms. The children will come to the health centre on days 0, 1, 2, 3, 7, 14, 21, 28, 35 and 42. If a child is not seen at the health centre he/she will be visited at home.

   6. Data Management The principle investigator will ensure that the study protocol is strictly adhered to and that data are correctly collected and recorded on the case record form. Data will be entered into an EpiData database during the study.

   7. Sample size The PCR corrected day 42 ACPR of AL was 97% in 2008 ( = before the national recommendation was changed in favour of A). It is likely that DP should be as efficacious as AL and it is therefore appropriate to conduct a non-inferiority trial13. Assuming 97% ACPR for both treatments, 5% significance level (alpha), 80% power (1-beta) and a non-inferiority limit (d) of 5% 144 children are required in each arm. Assuming a 20% loss to follow up a total of 346 children should be included.

   Analysis of data The data will be analysed using survival estimates of per protocol treatment failure rates but also intention to treat treatment failure rates. Final analysis will include a description of included children, proportions of adverse events and any serious adverse events, the proportion of children withdrawn or lost to follow up, the cumulative PCR corrected and uncorrected success and failure rates on day 42 and the proportion of early, late clinical and late parasitological treatment failures.

ELIGIBILITY:
Inclusion Criteria:

A) Age ≥6 months, and <13 years. B) Mono-infection with P. falciparum detected by microscopy. C) Parasitemia of 1.000-200.000/µl asexual forms. D) Axillary temperature ≥37.5 ˚C or a history of fever within 24 hours. E) Ability to swallow oral medication.

F) Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule. G) Informed consent from a parent or guardian

-

Exclusion Criteria:

A) Signs or symptoms of severe malaria, incl. hyperparasitaemia (>200.000/ µl asexual forms) B) Presence of general danger signs in children under 5 C) Presence of severe malnutrition. D) Any evidence of chronic disease or acute infection other than malaria. E) Regular medication which may interfere with antimalarial pharmacokinetics. F) History of hypersensitivity reactions or contraindications to AL, DP or quinine.

G) Domicile outside the study area.

-

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 346 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response rate | 42 days
  The data will be analysed using survival estimates of per protocol treatment failure rates but also intention to treat treatment failure rates.

SECONDARY OUTCOMES:
the safety of AL and DP | 42 days
  Self-reported signs and symptoms, clinical evaluations during treatment, day 7 and then weekly until day 42. leucocytes day 0, 3, 7, 14 and 21.

OTHER OUTCOMES:
To determine the capacity of each drug combination to protect against re-infection and to differentiate recrudescence from re-infections using PCR based methods | 42 days
Genetic polymorphisms in P. falciparum causing reparasitaemia (by PCR) and in 50 children perform a characterisation of P. falciparum geno- and phenotypes. | 42 days
  For all children with re-parasitaemia genetic polymorfisms will be established by PCR, and in additional 50 children further characterisation using cultures will be done
haemoglobin values | days 0, 3 and 42

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Jovel IT, Kofoed PE, Rombo L, Rodrigues A, Ursing J. Temporal and seasonal changes of genetic polymorphisms associated with altered drug susceptibility to chloroquine, lumefantrine, and quinine in Guinea-Bissau between 2003 and 2012. Antimicrob Agents Chemother. 2015 Feb;59(2):872-9. doi: 10.1128/AAC.03554-14. Epub 2014 Nov 24. PMID 25421474